CLINICAL TRIAL: NCT01771939
Title: Morphologic and Functional Results After Phacoemulsification and 25 Gauge Vitrectomy Versus Phacoemulsification Only in Eyes Affected by Idiopathic Epiretinal Membranes
Brief Title: Phacoemulsification and 25 Gauge (25G) Vitrectomy Versus Phacoemulsification Only in Idiopathic Epiretinal Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Marco Dal Vecchio, MD, University of Turin, Italy
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTCMER2
Record Dates: First submitted 2012-12-13; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Epiretinal Membrane
Keywords: Idiopathic epiretinal membranes; 25-G surgery in idiopathic epiretinal membranes
MeSH Terms: conditions — Epiretinal Membrane | interventions — Vitrectomy; Phacoemulsification; Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- idiopathic epiretinal membranes (Experimental): Patients in first arm, with worse visual condition, treated with 25-G Vitrectomy and phacoemulsification (cataract intervention)
  Interventions: Procedure: 25-G vitrectomy and phacoemulsification
- idiopathic epiretinal membrane (Active Comparator): Patient in second arm, with better pre-operative condition, treated with phacoemulsification (cataract intervention) only
  Interventions: Procedure: phacoemulsification (cataract surgery)

INTERVENTIONS:
Procedure: 25-G vitrectomy and phacoemulsification — 25-G vitrectomy with Internal Limiting Membrane peeling and phacoemulsification (cataract intervention)
  Arms: idiopathic epiretinal membranes
Procedure: phacoemulsification (cataract surgery) — lens extraction after phacoemulsification and intra-ocular artificial lens implantation
  Arms: idiopathic epiretinal membrane

SUMMARY:
The purpose of the study is to evaluate the difference in Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity, oct retinal thickness and microperimetry in 2 groups of 30 eyes each affected by idiopathic epiretinal membranes that underwent phacoemulsification and 25G pars-plana vitrectomy with internal limiting membrane (ILM) peeling (Group 1) versus phacoemulsification only (Group 2), with a follow-up length up to 5 years.

DETAILED DESCRIPTION:
Idiopathic epiretinal membranes represent a common cause of visual loss in elderly population. Vitrectomy with membrane peeling is nowadays considered the gold standard in the management of such pathology, with very good results either at short-time or at long-time follow up. In case of mild visual impairment due to epiretinal membrane and associated cataract, it is reasonable to treat only the lens pathology (with phacoemulsification and intra-ocular lens (IOL) implantation). In case of symptoms or ophthalmoscopic finding worsening it is always possible to submit patients who only underwent cataract surgery to vitrectomy with membrane peeling. There are, by now, no comparative studies between these two different approaches in medical literature.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic epiretinal membranes symptomatic

Exclusion Criteria:

* Absence of ocular symptoms, previous retinal interventions

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2006-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Visual acuity (using LogMar scale) changes from baseline to pre-defined periods after surgery | within 90,180,360,1360 days after surgery
  We observed how did the visual acuity (using LogMar scale) increase after the two different surgical approaches described.

SECONDARY OUTCOMES:
Microperimetry parameters and average macular thickness changes | within 90,180,360,1360 days after surgery
  We evaluated average sensitivity (SM) and local defect (DL) using microperimetry. We also evaluated the average macular thickness using optical coherence tomography technology.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Dal Vecchio, MD, Principal Investigator — Clinica Oculistica dell'Università, Ospedale Oftalmico Turin, Italy 10100; Antonio M. Fea, MD, PhD, Study Chair — Clinica Oculistica dell'Università, Ospedale Oftalmico Turin, Italy; Carlo A Lavia, MD, Principal Investigator — Clinica Oculistica dell'Università, Ospedale Oftalmico Turin, Italy
Locations (1):
- Clinica Oculistica dell'Università, Ospedale Oftalmico, Turin, Italy